CLINICAL TRIAL: NCT01943838
Title: A Phase 1 Dose-escalation Study of the Safety and Pharmacokinetics of a Tablet Formulation of SAR245408 Polymorph E Administered Once Daily to Subjects With Solid Tumors or Lymphoma
Brief Title: A Study of the Safety and Pharmacokinetics of SAR245408 Tablets in Patients With Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED12863; 2012-003368-39 (EudraCT Number); U1111-1132-9056 (Other: UTN)
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Neoplasm Malignant
MeSH Terms: conditions — Neoplasms | interventions — XL147

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SAR245408 polymorph E tablets (Experimental): Escalating doses of SAR245408 polymorph E tablets, once daily dosing with morning meal every day for two 28-days cycles
  Interventions: Drug: SAR245408

INTERVENTIONS:
Drug: SAR245408 — Pharmaceutical form: tablet Route of administration: oral

SUMMARY:
Primary Objective:

- To assess the safety, tolerability and plasma pharmacokinetics (PK) of SAR245408 given once daily as a tablet formulation of polymorph E in subjects with solid tumors or lymphoma.

DETAILED DESCRIPTION:
Screening: 1 to 28 days Study treatment period: two 28-day cycles (56 days) End-of-treatment visit: no later than 7 days after the last study drug administration Subjects not eligible for treatment continuation after Cycle 2 will be followed up for safety; a follow-up visit will be performed within 30 ± 3 days after the last study drug administration Subjects eligible for treatment continuation after Cycle 2 will be offered the opportunity to enroll in the treatment-extension study TED12414.

Total duration of study participation for each patient: 58 to 118 days.

ELIGIBILITY:
Inclusion criteria :

* Solid tumor that is metastatic or unresectable, or relapsed or refractory lymphoma (including chronic lymphocytic leukemia/small lymphocytic lymphoma), for which standard therapies are no longer effective or there are no therapies known to prolong survival or patient cannot tolerate or has contra-indication for a standard therapy and there is no alternative therapies.
* Male or female patient > or = 18 years old.
* Weight > or = 40 kg.
* Eastern Cooperative Oncology Group performance status < or = 1.
* Adequate white blood cells, platelets, and haemoglobin.
* Adequate liver and kidney functions.
* Fasting plasma glucose < 8.9 mmol/L.
* Sexually active patients using adequate contraception.
* Women of child-bearing potential with negative pregnancy test.

Exclusion criteria:

* Lymphoma involving the gastrointestinal tract.
* Prior treatment with cytotoxic chemotherapy (including investigational agents) or biologic agents (antibodies, immune modulators, and cytokines) within 4 weeks, or nitrosoureas or mitomycin C within 6 weeks, before the first dose of study drug.
* Prior treatment with a small-molecule kinase inhibitor (including investigational agents) within 2 weeks, or 5 half lives of the drug or active metabolites, whichever is longer, before the first dose of study drug.
* Any other investigational therapy within 4 weeks before the first dose of study drug.
* Intolerance to prior treatment with a PI3K inhibitor.
* Prior anticancer hormonal therapy within 2 weeks before the first dose of study drug.
* Prior radiation therapy within 2 weeks before the first dose of study drug.
* Uncontrolled brain metastases or primary brain tumor.
* Hereditary or acquired immunodeficiency syndrome or human immunodeficiency virus (HIV) infection.
* Positive serologies for Hepatitis B surface antigen (HBsAg) or anti-Hepatitis C virus (anti-HCV) antibodies.
* Patient is pregnant or breastfeeding.
* History of gastrointestinal surgery, or presence of gastrointestinal abnormality or disease, that may affect the pharmacokinetics of study drug.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities | Up to Day 28

SECONDARY OUTCOMES:
Number of patients with treatment-emergent adverse events | From first dose of SAR245408 up to 30 days after the last dose
Maximum SAR245408 plasma concentration | Days 1, 2, 8, 15, 29 and 30
Area under the SAR245408 plasma concentration versus time curve | Days 1, 2, 8, 15, 29 and 30

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 056001, Leuven, Belgium